CLINICAL TRIAL: NCT00108862
Title: A Strategy Study of Immediate Versus Deferred Initiation of Antiretroviral Therapy for AIDS Disease-Free Survival in HIV-Infected Persons Treated for Tuberculosis With CD4 Less Than 250 Cells/mm^3
Brief Title: Immediate Versus Deferred Start of Anti-HIV Therapy in HIV-Infected Adults Being Treated for Tuberculosis
Acronym: STRIDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5221; 1U01AI068636 (NIH); ACTG A5221 (Other: AIDS Clinical Trials Group)
Record Dates: First submitted 2005-04-19; First posted 2005-04-20 (Estimated); Results first posted 2011-11-02 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: HIV Infection; Tuberculosis
Keywords: Treatment Naive; TB; HIV; Antiretroviral Agents; Strategy Study
MeSH Terms: conditions — HIV Infections; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate ART (Experimental): The intervention is the strategy of initiating antiretroviral therapy (ART) after approximately 2 weeks of tuberculosis (TB) treatment.
  Interventions: Other: Strategy: Immediate ART
- Deferred ART (Active Comparator): The intervention is the strategy of initiating ART after 8 to 12 weeks of TB treatment.
  Interventions: Other: Strategy: Deferred ART

INTERVENTIONS:
Other: Strategy: Immediate ART — The intervention is the strategy of initiating antiretroviral therapy (ART) after approximately 2 weeks of rifampin (RIF)- or other rifamycin-based TB treatment according to in-country national TB treatment guidelines. The study-provided ART is efavirenz (EFV) 600 mg (1 tablet orally), emtricitabine (FTC) 200 mg (1 capsule orally), and tenofovir disoproxil fumarate (TDF) 300 mg (1 tablet orally) daily. Substitutions with other locally available U.S. Food and Drug Administration (FDA)-approved or tentatively approved antiretrovirals that are compatible with TB treatment may be used at the discretion of the site investigator. The TB treatment will be supplied and monitored by the host country TB control program.
  Arms: Immediate ART
Other: Strategy: Deferred ART — The intervention is the strategy of initiating ART either after 8-12 weeks of RIF- or other rifamycin-based TB treatment according to in-country national TB treatment guidelines. The study-provided ART is EFV 600 mg (1 tablet orally), FTC 200 mg (1 capsule orally), and TDF 300 mg (1 tablet orally) daily. Initiation outside of these windows, on a case by case basis, is permitted at the discretion of the site investigator. Substitutions with other locally available U.S. FDA-approved or tentatively approved antiretrovirals that are compatible with TB treatment may be used at the discretion of the site investigator. The TB treatment will be supplied and monitored by the host country TB control program.
  Other Names: Early ART
  Arms: Deferred ART

SUMMARY:
The purpose of this study is to determine the best time to begin anti-HIV treatment in individuals who have HIV and tuberculosis (TB).

Study hypothesis: Immediate antiretroviral therapy (ART), initiated after approximately 2 weeks of TB treatment, will reduce the frequency of other AIDS-defining illnesses and death in HIV-infected participants being treated for TB by at least 40% at week 48 when compared to deferred ART, initiated at after 8-12 weeks of TB treatment.

DETAILED DESCRIPTION:
Tuberculosis (TB) is the most important co-infection in the HIV epidemic; the bi-directional relationship between the two diseases is well established. HIV increases the risk for TB acquisition, reactivation, and reinfection, and reduces survival compared to patients with TB alone. In individuals with HIV, TB infection results in reduced survival, increased risk for opportunistic infections, and elevations in HIV replication. Improving the outcome of HIV-infected individuals who develop TB is of high importance. Initiating antiretroviral therapy (ART) shortly after initiating TB treatment may improve outcomes in individuals co-infected with HIV and TB. However, data to support this suggestion were limited before this study began. This study will determine the most appropriate time to initiate ART in HIV-infected individuals who recently initiated treatment for TB.

This study lasted 48 weeks and comprised two steps. At study entry, participants underwent clinical assessment, drug adherence training, and blood collection. In Step 1, participants were randomly assigned to one of two arms. Participants in Arm A initiated ART after approximately 2 weeks of TB treatment. Participants in Arm B deferred ART until after 8 to 12 weeks of TB treatment. In Step 2, Arm B participants initiated ART; Arm A participants did not enter Step 2. ART consisted of efavirenz (EFV) and emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF); FTC and TDF could be given as individual agents. Drug substitutions could be made for participants who could not tolerate the specified regimen. Blood collection and clinical assessments occurred at weeks 4, 8, 12, 16, 24, 32, 40, and 48.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected.
* Confirmed or probable TB (more information on the criterion can be found in the protocol).
* Chest x-ray within 30 days prior to study entry.
* Receipt of 1-14 cumulative days of rifampin- or other rifamycin-based TB treatment that was initiated within 28 days prior to study entry.
* CD4 count less than 250 cells/mm^3 within 30 days prior to study entry.
* Willing to use acceptable methods of contraception while on study drugs and for 6 weeks after stopping these drugs.
* Able to swallow oral medications.
* Parent of guardian willing to provide informed consent, if applicable.
* Karnofsky performance score =>20 at time of study entry.

Exclusion Criteria:

* ART for longer than 7 cumulative days prior to study entry or treatment for any period of time with one or more antiretrovirals. Participants who have taken ART during pregnancy or for occupational exposure are not excluded.
* Allergy or sensitivity to any of the study drugs or their formulations.
* History of multidrug-resistant TB.
* Receipt of any investigational therapy or chemotherapy within 30 days prior to study entry.
* Certain medications.
* Breastfeeding.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 809 (Actual)
Dates: Start 2006-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Havlir, MD, Study Chair — San Francisco General Hospital and University of California, San Francisco
Locations (26):
- United States (4):
  - University of Southern California (1201), Los Angeles, California
  - University of California, San Diego, AVRC CRS (701), San Diego, California
  - University of California, San Francisco AIDS CRS (801), San Francisco, California
  - NY Univ. HIV/AIDS CRS (401), New York, New York
- Botswana (2):
  - Gaborone Prevention/Treatment Trials CRS (12701), Gaborone
  - Molepolole Prevention/Treatment Trials CRS (12702), Molepolole
- Brazil (3):
  - Hospital Nossa Senhora da Conceicao CRS (12201), Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa Clinica Evandro Chagas (12101), Rio de Janeiro
  - Projecto Praca Onze/Hesfa CRS (30333), Rio de Janeiro
- Les Centres GHESKIO CRS (30022), Bicentenaire, Port-au-Prince, Haiti
- India (2):
  - National AIDS Research Institute Pune CRS (11601), Pune, Maharashtra
  - Y.R.G Ctr, for AIDS Research and Education (11701), Chennai
- Kenya (2):
  - AMPATH at Moi Univ. Teaching Hosp. Eldoret CRS (12601), Eldoret
  - Walter Reed Project - Kenya Med. Research Institute Kericho CRS (12501), Kericho
- Malawi (2):
  - College of Med. JHU CRS (30301), Blantyre
  - University of North Carolina Lilongwe CRS (12001), Lilongwe
- Peru (2):
  - Investigaciones Medicas en Salud (INMENSA) (11302), San Isidro, Lima region
  - Asociacion Civil Impacta Salud y Educacion - Miraf CRS (11301), Lima
- South Africa (4):
  - CAPRISA eThekwini CRS (31422), Durban, KwaZulu-Natal
  - Durban Adult HIV CRS (11201), Durban
  - Soweto ACTG CRS (12301), Johannesburg
  - Univ. of Witwatersrand CRS (11101), Johannesburg
- Chiang Mai University ACTG CRS (11501), Chiang Mai, Thailand
- Joint Clinical Research Centre (JCRC) (12401), Kampala, Uganda
- Kalingalinga Clinic CRS (12801), Lusaka, Zambia
- UZ-Parirenyatwa CRS (30313), Harare, Zimbabwe

REFERENCES:
- [Derived] Crump JA, Wu X, Kendall MA, Ive PD, Kumwenda JJ, Grinsztejn B, Jentsch U, Swindells S. Predictors and outcomes of Mycobacterium tuberculosis bacteremia among patients with HIV and tuberculosis co-infection enrolled in the ACTG A5221 STRIDE study. BMC Infect Dis. 2015 Jan 13;15:12. doi: 10.1186/s12879-014-0735-5. PMID 25582793
- [Derived] Havlir DV, Kendall MA, Ive P, Kumwenda J, Swindells S, Qasba SS, Luetkemeyer AF, Hogg E, Rooney JF, Wu X, Hosseinipour MC, Lalloo U, Veloso VG, Some FF, Kumarasamy N, Padayatchi N, Santos BR, Reid S, Hakim J, Mohapi L, Mugyenyi P, Sanchez J, Lama JR, Pape JW, Sanchez A, Asmelash A, Moko E, Sawe F, Andersen J, Sanne I; AIDS Clinical Trials Group Study A5221. Timing of antiretroviral therapy for HIV-1 infection and tuberculosis. N Engl J Med. 2011 Oct 20;365(16):1482-91. doi: 10.1056/NEJMoa1013607. PMID 22010914

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited at 26 sites from 13 countries: 4 each from U.S. and South Africa; 3 from Brazil; 2 each from Peru, Botswana, Kenya, Malawi, and India; and 1 each from Haiti, Uganda, Zambia, Zimbabwe, and Thailand, between September 2006 and August 2009.
Pre-assignment Details: HIV-infected persons at least 13 years of age, naive to antiretroviral therapy, who had received 1-14 cumulative days of a rifamycin-based TB regimen within 28 days prior to study entry, and had a CD4 count <250 cells/mm3. Randomization was stratified by screening CD4 (<50 vs =>50). Three participants were deemed ineligible and taken off study.
Groups:
- Immediate ART: These participants initiated HIV antiretroviral therapy (ART) within 72 hours of randomization, which took place at most 2 weeks after initiating rifampin (RIF)- or other rifamycin-based TB treatment according to in-country national TB treatment guidelines. The study-provided drugs were efavirenz (EFV) 600 mg (provided to non-U.S. sites only; 1 tablet orally) and emtricitabine (FTC) 200 mg/tenofovir disoproxil fumarate (TDF) 300 mg (1 fixed-dose combination tablet orally) once daily. FTC 200 mg (1 capsule) and TDF 300 mg (1 tablet) could be substituted for the fixed-dose combination tablet and was provided by the study. Participants who could not tolerate EFV could be offered nevirapine (NVP) 200 mg daily for 14 days, then 200 mg twice daily. Substitutions with other locally-available U.S. Food and Drug Administration (FDA)-approved or tentatively approved antiretrovirals (ARVs) that were compatible with TB therapy could be used at the discretion of the site investigator.
- Deferred ART: These participants deferred ART until 8 to 12 weeks after initiation of their RIF- or other rifamycin-based TB treatment according to in-country national TB treatment guidelines. The study-provided drugs were EFV 600 mg (provided to non-U.S. sites only; 1 tablet orally) and FTC 200 mg/TDF 300 mg (1 fixed-dose combination tablet orally) once daily. FTC 200 mg (1 capsule) and TDF 300 mg (1 tablet) could be substituted for the fixed-dose combination tablet and was provided by the study. Participants who could not tolerate EFV could be offered NVP 200 mg daily for 14 days, then 200 mg twice daily. Substitutions with other locally-available U.S. FDA-approved or tentatively approved ARVs that were compatible with TB therapy could be used at the discretion of the site investigator.
Period: Overall Study
Arm/Group | Immediate ART | Deferred ART
Started | 405 | 401 (Three participants who were deemed clinically ineligible and taken off study were omitted.)
Completed | 337 | 339
Not Completed | 68 | 62
Not completed — Death | 31 | 37
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Lost to Follow-up | 27 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate ART | Deferred ART | Total
Number analyzed (Participants) | 405 | 401 | 806
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 403 | 398 | 801
  >=65 years | 2 | 1 | 3
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [29 to 40] | 34 [29 to 42] | 34 [29 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 166 | 305
  Male | 266 | 235 | 501
Region of Enrollment [Number; unit: participants]
  South Africa | 109 | 112 | 221
  Malawi | 69 | 68 | 137
  Brazil | 57 | 56 | 113
  Kenya | 36 | 36 | 72
  Peru | 23 | 25 | 48
  India | 26 | 21 | 47
  Zambia | 17 | 17 | 34
  Zimbabwe | 16 | 17 | 33
  Uganda | 15 | 14 | 29
  Botswana | 13 | 15 | 28
  Haiti | 12 | 8 | 20
  United States | 9 | 10 | 19
  Thailand | 3 | 2 | 5
TB Diagnosis Level at Entry [Number; unit: participants]
  Confirmed TB | 193 | 181 | 374
  Probable TB | 208 | 218 | 426
  Not TB | 4 | 2 | 6
Drug-Resistant TB Status at Entry [Number; unit: participants]
  Rifampin (RIF) Resistant TB | 1 | 0 | 1
  Isoniazid (INH) Resistant TB | 3 | 5 | 8
  RIF and INH Resistant TB (Multi-Drug Resistant TB) | 1 | 4 | 5
  RIF and INH Sensitive TB | 400 | 392 | 792
Time to ART Start from Start of TB Medications [Median (Inter-Quartile Range); unit: days] | 10 [7 to 12] | 70 [66 to 75] | 14 [10 to 70]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Survived Without AIDS Progression.
Description: As this was a study of the strategy of providing antiretroviral therapy (ART) during the initial treatment of TB versus deferring ART until TB was treated for 8-12 weeks, all eligible participants randomized were followed for 48 weeks, whether they started ART as scheduled, whether they started ART at all, or even if the participant did not have TB and discontinued TB treatment. The percent surviving without a new AIDS-defining illness was calculated using a Kaplan-Meier estimator with an associated standard error.
Time Frame: Through week 48
Population: Numbers presented use the intent-to-treat approach (i.e., ignoring changes from randomized treatment strategy).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Immediate ART | Deferred ART
Number analyzed (Participants) | 405 | 401
percent of participants | 13 [10 to 16] | 16 [12 to 20]
Statistical Analysis 1: Comparison: Immediate ART vs Deferred ART; Assuming that immediate ART was better than deferred ART and that the combined rate in the deferred ART arm was 25% compared to 15% in the immediate ART arm (a 40% reduction), and assuming 10% loss to follow-up in a two-sided, two-sample 0.05-level asymptotically-normal test with 400 participants in each arm, there was 90% power. The percents tested were Kaplan-Meier estimators at week 48 with the associated Greenwood's variance; Test type: Superiority or Other; p = 0.45, Z-test, 2-sided — The analysis was stratified by screening CD4 (<50 cells/mm3 vs =>50). Interim reviews employed group sequential monitoring using an O'Brien-Fleming use function. At final analysis, the a priori threshold for statistical significance was 0.0492; A 2-sided Z-test was used to compare the two percents. The test was weighted by the inverse of the Greenwood's variance in each CD4 stratum; Mean Difference (Final Values) = 3, 95.08% CI 2-sided [-2 to 8], Standard Error of Mean 3 — The difference in percents was calculated as the percent failed in the Deferred ART arm minus the percent failed in the Immediate ART arm

2. Other Pre Specified Outcome: Percent of Participants in the Less Than 50 Cells/mm^3 CD4 Stratum Who Survived Without AIDS Progression.
Description: Participants were included as described in the Outcome Measure Description for the Primary Outcome, except that only those in the <50 CD4 stratum were analyzed. The percent surviving without a new AIDS-defining illness was calculated using a Kaplan-Meier estimator with an associated standard error.
Time Frame: Through week 48
Population: Numbers presented use the intent-to-treat approach (i.e., ignoring changes from randomized treatment strategy).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Immediate ART | Deferred ART
Number analyzed (Participants) | 144 | 141
percent of participants | 16 [10 to 21] | 27 [19 to 39]
Statistical Analysis 1: Comparison: Immediate ART vs Deferred ART; The study was not powered for this pre-specified subgroup analysis; Test type: Superiority or Other; p = 0.02, Z-test, 2-sided — Interim reviews employed group sequential monitoring using an> O'Brien-Fleming use function. At final analysis, the a priori threshold for statistical significance was 0.0492; Mean Difference (Final Values) = 11, 95.08% CI 2-sided [2 to 21], Standard Error of Mean 5 — [estimate comment as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Percent of Participants in the Greater Than or Equal to 50 Cells/mm^3 CD4 Stratum Who Survived Without AIDS Progression.
Description: Participants were included as described in the Outcome Measure Description for the Primary Outcome, except that only those in the =>50 CD4 stratum were analyzed. The percent surviving without a new AIDS-defining illness was calculated using a Kaplan-Meier estimator with an associated standard error.
Time Frame: Through week 48
Population: Numbers presented use the intent-to-treat approach (i.e., ignoring changes from randomized treatment strategy).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Immediate ART | Deferred ART
Number analyzed (Participants) | 261 | 260
percent of participants | 11 [8 to 15] | 10 [7 to 14]
Statistical Analysis 1: Comparison: Immediate ART vs Deferred ART; The study was not powered for this pre-specified subgroup analysis; Test type: Superiority or Other; p = 0.67, Z-test, 2-sided — Interim reviews employed group sequential monitoring using an O'Brien-Fleming use function. At final analysis, the a priori threshold for statistical significance was 0.0492; Mean Difference (Final Values) = -1, 95.08% CI 2-sided [-7 to 4], Standard Error of Mean 3 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percent of Participants Reporting a Grade 3 or 4 Adverse Event or Laboratory Abnormality
Description: All eligible participants were included in this analysis. The percent of participants whose highest reported grade of adverse events and laboratory abnormalities was Grade 3 or 4 was calculated with an associated standard error, where Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening/disabling, and Grade 5=death.
Time Frame: Through week 48
Population: Numbers presented use the intent-to-treat approach (i.e., ignoring changes from randomized treatment strategy).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Immediate ART | Deferred ART
Number analyzed (Participants) | 405 | 401
percent of participants | 44 [39 to 49] | 47 [42 to 52]

5. Secondary Outcome: Time to First New AIDS-defining Illness or Death.
Description: All eligible participants were included in this analysis. Weeks from randomization to first new AIDS-defining illness or death was analyzed using a stratified Cox proportional hazards regression model. The stratification was by screening CD4 cell count: <50 cells/mm3 versus =>50 cells/mm3.
Time Frame: Through week 48
Population: Numbers presented use the intent-to-treat approach (i.e., ignoring changes from randomized treatment strategy).
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Immediate ART | Deferred ART
Number analyzed (Participants) | 405 | 401
weeks
  5th percentile | 4 [3 to 8] | 7 [4 to 10]
  10th percentile | 13 [8 to 49] | 12 [9 to 19]

6. Secondary Outcome: Percent of Participants With Culture-confirmed Tuberculosis (TB) Who Survived Without AIDS Progression.
Description: This analysis was based on 374 participants with culture-confirmed TB at entry. The percent with culture-confirmed TB surviving without a new AIDS-defining illness was calculated using a Kaplan-Meier estimator with an associated standard error.
Time Frame: Through week 48
Population: Numbers presented use the intent-to-treat approach (i.e., ignoring changes from randomized treatment strategy).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Immediate ART | Deferred ART
Number analyzed (Participants) | 193 | 181
percent of participants | 12 [7 to 17] | 17 [12 to 23]

7. Secondary Outcome: Percent of Participants Who Interrupted or Discontinued at Least One Tuberculosis (TB) Medication Due to Toxicity.
Description: All eligible participants were included in this analysis. The percent of participants who interrupted at least one TB medication for more than one day due to toxicity or discontinued at least one TB medication due to toxicity was calculated with an associated standard error.
Time Frame: Through week 48
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Immediate ART | Deferred ART
Number analyzed (Participants) | 405 | 401
percent of participants | 9 [6 to 12] | 10 [7 to 13]

8. Secondary Outcome: Percent of Participants With Confirmed or Probable Tuberculosis (TB) Whose TB Resolved, or Who Required TB Treatment Through the End of Follow-up, or Died, or Were Lost to Follow-up.
Description: TB treatment outcome was assessed in the 800 eligible participants who had confirmed or probable TB at study entry. The sites determined if the TB was resolved. If TB was not resolved, TB treatment outcome status was determined based on whether TB treatment was ongoing at the last study visit; if the participant died while TB treatment was ongoing; or if the participant was lost to follow-up, withdrew consent, or other reason for lacking TB resolution status. Percents were calculated with associated standard errors.
Time Frame: Through week 48
Population: Participants with confirmed or probable TB at study entry were included in this analysis. Numbers presented use the intent-to-treat approach (i.e., ignoring changes from randomized treatment strategy).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Immediate ART | Deferred ART
Number analyzed (Participants) | 401 | 399
percent of participants
  TB Resolved | 79 [75 to 83] | 82 [78 to 85]
  TB Treatment Ongoing | 6 [4 to 9] | 5 [3 to 8]
  Death | 6 [4 to 9] | 7 [5 to 10]
  Lost-to-Follow-up/Withdrew Consent/Other | 8 [5 to 11] | 6 [4 to 9]

9. Secondary Outcome: Percent of Participants Whose CD4 Increased by at Least 100 Cells/mm^3 Between Baseline and Week 48.
Description: All eligible participants were included in the analysis. Participants who were lost-to-follow-up (LFU) prior to week 48 or who were alive with a CD4 cell count increase of less than 100 cells/mm^3 were grouped separately those who died or whose CD4 cell count increased by at least 100 cells/mm^3. Participants missing CD4 cell counts at week 48 were coded as LFU in this analysis. The percents were calculated with associated standard errors.
Time Frame: Through week 48
Population: Numbers presented use the intent-to-treat approach (i.e., ignoring changes from randomized treatment strategy).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Immediate ART | Deferred ART
Number analyzed (Participants) | 405 | 401
percent of participants
  CD4 increase of at least 100 cells/mm^3 | 60 [55 to 65] | 60 [55 to 65]
  LFU, or alive with CD4 increase < 100 cells/mm^3 | 32 [28 to 37] | 31 [26 to 35]
  Dead | 8 [5 to 11] | 9 [7 to 13]

10. Secondary Outcome: Percent of Participants With MTB IRIS.
Description: All eligible participants were included in this analysis. The percent of participants with Mycobacteria tuberculosis (MTB)-associated immune reconstitution inflammatory syndrome (IRIS) was calculated with an associated standard error.
Time Frame: Through week 48
Population: Numbers presented use the intent-to-treat approach (i.e., ignoring changes from randomized treatment strategy).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Immediate ART | Deferred ART
Number analyzed (Participants) | 405 | 401
percent of participants | 11 [8 to 14] | 5 [3 to 7]

11. Secondary Outcome: Percent of Participants With HIV IRIS.
Description: All eligible participants were included in this analysis. The percent of participants with HIV-associated immune reconstitution inflammatory syndrome (IRIS) was calculated with an associated standard error.
Time Frame: Through week 48
Population: Numbers presented use the intent-to-treat approach (i.e., ignoring changes from randomized treatment strategy).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Immediate ART | Deferred ART
Number analyzed (Participants) | 405 | 401
percent of participants | 3 [2 to 5] | 3 [1 to 5]

12. Secondary Outcome: Percent of Participants Whose HIV Viral Load Was Less Than 400 Copies/mL at Week 48.
Description: All eligible participants were included in the analysis. Participants who were lost-to-follow-up (LFU) prior to week 48 or who were alive with a HIV viral load at least 400 copies/mL were grouped separately those those who died or who had HIV viral loads below 400 copies/mL. Participants missing HIV viral loads at week 48 were coded as LFU in this analysis. Percents were calculated with associated standard errors.
Time Frame: Through week 48
Population: Numbers presented use the intent-to-treat approach (i.e., ignoring changes from randomized treatment strategy).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Immediate ART | Deferred ART
Number analyzed (Participants) | 405 | 401
percent of participants
  HIV viral load < 400 copies/mL | 72 [68 to 77] | 75 [71 to 79]
  LFU, or alive with HIV viral load at least 400 | 20 [16 to 24] | 16 [12 to 20]
  Dead | 8 [5 to 11] | 9 [7 to 13]

ADVERSE EVENTS:
Time Frame: Through week 48
Arm/Group | Immediate ART | Deferred ART
Serious Adverse Events (participants affected / at risk) | 55/405 | 44/401
Other Adverse Events (participants affected / at risk) | 391/405 | 389/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate ART (N=405) | Deferred ART (N=401)
Anaemia (Blood and lymphatic system disorders) | 6 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 2 | 6
Pyrexia (General disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 2
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 5 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Meningitis bacterial (Infections and infestations) | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 0 | 3
Meningitis tuberculous (Infections and infestations) | 2 | 1
Mycobacterium avium complex infection (Infections and infestations) | 2 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 7 | 1
Sepsis (Infections and infestations) | 0 | 3
Tuberculoma of central nervous system (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Viral myocarditis (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system mass (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Coma hepatic (Nervous system disorders) | 1 | 0
Encephalitis (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 2
Renal impairment (Renal and urinary disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate ART (N=405) | Deferred ART (N=401)
Lymphadenopathy (Blood and lymphatic system disorders) | 37 | 19
Abdominal pain (Gastrointestinal disorders) | 27 | 21
Diarrhoea (Gastrointestinal disorders) | 23 | 33
Leukoplakia oral (Gastrointestinal disorders) | 20 | 30
Nausea (Gastrointestinal disorders) | 21 | 18
Vomiting (Gastrointestinal disorders) | 42 | 39
Chest pain (General disorders) | 26 | 20
Pyrexia (General disorders) | 75 | 63
Herpes zoster (Infections and infestations) | 19 | 22
Oral candidiasis (Infections and infestations) | 47 | 78
Pneumonia bacterial (Infections and infestations) | 29 | 34
Alanine aminotransferase increased (Investigations) | 79 | 82
Aspartate aminotransferase increased (Investigations) | 132 | 152
Blood albumin (Investigations) | 18 | 21
Blood albumin abnormal (Investigations) | 307 | 323
Blood alkaline phosphatase increased (Investigations) | 133 | 138
Blood bicarbonate abnormal (Investigations) | 78 | 89
Blood bilirubin increased (Investigations) | 26 | 27
Blood creatinine increased (Investigations) | 29 | 28
Blood phosphorus decreased (Investigations) | 71 | 56
Blood potassium decreased (Investigations) | 38 | 33
Blood sodium decreased (Investigations) | 212 | 227
Haemoglobin decreased (Investigations) | 211 | 215
Neutrophil count decreased (Investigations) | 86 | 102
Platelet count decreased (Investigations) | 19 | 34
Weight decreased (Investigations) | 21 | 16
White blood cell count decreased (Investigations) | 64 | 75
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 22
Dizziness (Nervous system disorders) | 33 | 31
Headache (Nervous system disorders) | 41 | 53
Cough (Respiratory, thoracic and mediastinal disorders) | 47 | 44
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 25
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 21 | 39
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 24
Rash (Skin and subcutaneous tissue disorders) | 35 | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.